CLINICAL TRIAL: NCT04252430
Title: Open Label, Phase I Study to Assess and Compare the Pharmacokinetic Parameters After Single Oral Administration of MD1003 100 mg in Renal Impaired Patients and Healthy Subjects With Normal Renal Function
Brief Title: RI Study to Assess and Compare the Pharmacokinetic Parameters of MD1003 in Renal Impaired Patients and Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to other phase 3 trial failure to meet primary endpoint
Sponsor: MedDay Pharmaceuticals SA (Industry)
Collaborators: Eurofins Optimed (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: MD1003CT2019602RI; 2019-002315-26 (EudraCT Number)
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2019-10

CONDITIONS: Healthy Volunteers; Impaired Renal Function
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: Open label, Parallel-group, Single oral dose
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with renal impaired function (Active Comparator): 6 patients with mild renal impaired function, 6 patients with moderate renal impaired function and 6 patients with severe ranal impaired function
  Interventions: Drug: MD1003
- Healthy subjects (Active Comparator): Healthy volunteers will be matched with impaired renal function patients
  Interventions: Drug: MD1003

INTERVENTIONS:
Drug: MD1003 — Single oral dose administration of MD1003 at Day 1

SUMMARY:
This is a Phase 1, multicentric, open-label,two arms to assess and compare the effect of single oral administration of MD1003 on the pharmacokinetic parameters in renal impaired patients and healthy subjects with normal renal function.

The planned enrollment is 36 subjects (18 impaired patients and 18 healthy subjects).

DETAILED DESCRIPTION:
The study is a multicentric, open label, phase I, two arms study to compare pharmacokinetics of MD1003 after a single oral dose of MD1003 100 mg in 18 healthy male volunteers and in 18 renal impaired patients.

It is planned to enroll a total of 36 subjects to receive a single oral dose of investigational medicinal product (IMP):

* 6 patients with mild renal impaired function, 6 patients with moderate renal impaired function and 6 patients with severe renal impaired function will be enrolled in four Hungarian centers;
* 18 Healthy volunteers will be enrolled by Eurofins Optimed in Gières, France. Healthy volunteers will be matched with impaired renal function patients on ethnic group, sex, age and BMI.

Subjects will be screened for eligibility to participate in the study up to 21 days prior to the first administration. For both arms, subjects will be admitted into the Clinical Research Unit (CRU) on Day -3. On the morning of Day 1, subjects will receive a single 100 mg oral dose of MD1003 following an overnight fast (i.e., at least 10 hours). Subjects will be confined to the CRU until discharge on Day 8 with PK blood sample draws for measurement of MD1003 and its main metabolites being taken throughout the confinement (Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose). Urine sample draws for measurement of MD1003 and its main metabolites will also be taken throughout the study (pre-dose, ]D1T0h - D1T4h], ]D1T4h - D1T8h], ]D1T8h - D1T12h], ]D1T12h - D2T24h], ]D2T24h - D2T36h], ]D2T36h - D3T48h], ]D3T48h - D4T72h], ]D4T72h - D5T96h], ]D5T96h - D6T120h], ]D6T120h - D7T144h], ]D7T144h - D8T168h] post-dose). Then, subjects will come back to the CRU for 4 ambulatory visits on Day 10, Day 12, Day 14 and Day 16 for blood sampling (respectively 216, 264, 312, 360 hours post dose).

A follow-up post study visit will occur on Day 23 (±2 days) post-dose to ensure the ongoing wellbeing of the subjects.

Adverse events (AEs), clinical laboratory evaluations, vital signs assessments, 12-lead ECG and physical examination (PE) findings will be monitored at screening and at specified times during the study. All AEs will be recorded throughout the study (i.e., from signing of the Informed Consent Form until Study Completion).

The Study Completion is defined as the last subject's end-of-study assessment.

ELIGIBILITY:
Inclusion Criteria:

For eligibility into the trial, subjects and patients must meet all the following inclusion criteria:

1. Male or female subjects, aged 18 to 75 years inclusive
2. Females participating in this study must be of non-childbearing potential or using highly effective contraception for the full duration of the study and for 1 month after the end of treatment, as described below:

   * Cessation of menses for at least 12 months due to ovarian failure;
   * Surgical sterilization such as bilateral oophorectomy, hysterectomy, or medically documented ovarian failure;
   * Using an highly effective non-hormonal method of contraception (bilateral tubal occlusion, vasectomized partner or intra-uterine device);
   * Double contraception with barrier AND highly effective hormonal method of contraception (oral, intravaginal or transdermal combined estrogen and progestogen hormonal contraception associated with inhibition of ovulation, oral, injectable or implantable progestogen-only hormonal contraception associated with inhibition of ovulation or intrauterine hormone-releasing system). The hormonal contraception must be started at least one month prior to inclusion.
3. Negative serum pregnancy test at screening (if applicable);
4. Normal hepatic function;
5. Non-smoker subject or smoker of not more than 5 cigarettes a day;
6. Signing a written informed consent prior to selection;
7. Covered by Health Insurance System and / or in compliance with the recommendations of National Law in force relating to biomedical research.

For renal impaired patients:

1. Renal impairment patients with mild decrease in estimated creatinine clearance (CLcr) (60 ≤ CLcr ≤ 89 mL.min) or with moderate decrease of CLcr (30 ≤ CLcr ≤ 59 mL.min) or severe decrease of CLcr (15 ≤ CLcr ≤ 29 mL.min) using the Cockcroft-Gault equation;
2. Supine blood pressure ≤ 170/110 mmHg;
3. Documented renal impairment indicated by reduced estimated creatinine clearance within 12 months of screening or longer;
4. Stable renal function as evidenced by ≤ 30% difference in two evaluation of estimated creatinine clearance on two separate occasions separated by at least 28 days with one measurement being the value at screening;
5. Body Mass Index (BMI) between 20 and 34 kg/m2 inclusive.

For healthy subjects with normal renal function:

1. Considered as healthy after a comprehensive clinical assessment (detailed medical history and complete physical examination);
2. Estimated creatinine clearance (CLcr) ≥ 90 mL/min;
3. No proteinuria (< 0.15 g/L determined by urinalysis);
4. Body Mass Index (BMI) between 20 and 30 kg/m2 inclusive and body weight (BW) not lower than 55 kg;
5. Normal Blood Pressure (BP) and Heart Rate (HR) at the screening visit after 10 minutes in supine position:

   * 90 mmHg ≤ Systolic Blood Pressure (SBP) ≤ 145 mmHg,
   * 50 mmHg ≤ Diastolic Blood Pressure (DBP) ≤ 90 mmHg,
   * 45 bpm ≤ HR ≤ 90 bpm,
   * Or considered NCs by investigators;
6. Normal ECG recording on a 12-lead ECG at the screening visit:

   * 120 < PR < 220 ms,
   * QRS < 110 ms,
   * QTcf ≤ 430 ms for male and < 450 ms for female,
   * No sign of any trouble of sinusal automatism,
   * Or considered NCs by investigators;
7. Laboratory parameters within the normal range of the laboratory (hematological, blood chemistry tests, urinalysis). Individual values out of the normal range can be accepted if judged clinically non relevant by the Investigator;
8. Normal dietary habits;
9. Matched to at least 1 renal impaired patient by ethnic group, sex, age (+/- 10 years) and BMI (+/- 20%).

Exclusion Criteria:

1. Positive Hepatitis B surface (HBs) antigen or anti Hepatitis C Virus (HCV) antibody, or positive results for Human Immunodeficiency Virus (HIV) 1 or 2 tests);
2. History or presence of drug or alcohol abuse (alcohol consumption > 40 grams/day);
3. Subject/Patient who, in the judgment of the Investigator, is likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language problem, poor mental development;
4. Subject/Patient who cannot be contacted in case of emergency;
5. History or presence of allergy or unusual reactions to some drugs or anesthetics or known hypersensitivity to the investigation product or its excipients (including lactose intolerance);
6. Any medications intake within 3 months that may interfere with absorption, distribution, metabolism or excretion of the study drug, or any medication that may result in induction or inhibition of microsomal enzymes;
7. Subject/Patient who is in the exclusion period of a previous study;
8. Administrative or legal supervision;
9. Blood donation (including in the frame of a clinical trial) within 2 months before administration or blood donation planned during the study or within 2 months following participation to the study;
10. Subject/Patient who is pregnant or breastfeeding. Subject/Patient should not be enrolled if she plans to become pregnant during the time of study participation;
11. Excessive consumption of beverages with xanthine bases (> 4 cups or glasses / day);
12. Positive results of screening for drugs of abuse;
13. Intake of any food or any beverage containing grapefruit or grapefruit juice within 48h prior to the first dosing and the inability to stop such intake during the study;
14. Evidence or history of clinically significant uncontrolled hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, metabolic, systemic, infectious, or allergic disease (including drug hypersensitivity or allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing);
15. General anesthesia within 3 months before administration;
16. Major surgery within 28 days prior to inclusion or major surgery planned during the next 6 months.

For renal impaired patients:

1. History of renal transplant;
2. The patient has evidence of an unstable clinically important medical condition other than impaired renal function;
3. The patient has an acute exacerbation or unstable renal function, as indicated by worsening of clinical and/or laboratory signs of renal impairment, within the 4 weeks before study drug administration;
4. Patients undergoing any method of dialysis or hemofiltration;
5. Disorders or surgery of the gastrointestinal tract which may interfere with drug absorption or may otherwise influence the pharmacokinetics of the investigational medicinal product (e.g., inflammatory bowel disease, resections of the small or large intestine, etc.);
6. History of febrile illness within 5 days prior to dosing;
7. Evidence of clinically significant liver disease or liver damage (e.g., hepatitis B or C, autoimmune hepatitis, primary biliary cirrhosis, non-alcoholic fatty liver disease, elevated aspartate aminotransferase (AST) or alanine aminotransferase (ALT) that is considered clinically significant by the Investigator, etc.). Presence or history of protein drug hypersensitivity, or allergic disease diagnosed and treated by a physician;
8. Any drug intake during the 2 weeks or 5 half-lives of the drug preceding the first administration.

For Healthy subjects with normal renal function:

1. Any history or presence of renal disease
2. Frequent headaches (> twice a month) and / or migraines, recurrent nausea and / or vomiting;
3. Symptomatic hypotension whatever the decrease of blood pressure or asymptomatic postural hypotension defined by a decrease in SBP (≥20 mmHg) or DBP (≥20 mmHg) within two minutes when changing from the supine to the standing position;
4. Inability to abstain from intensive muscular effort;
5. Any drug intake (except paracetamol 3g/d or contraception) during the 2 weeks or 5 half-lives of the drug preceding the first administration;
6. Subject who would receive more than 4500 euros as indemnities for his participation in biomedical research within the 12 last months, including the indemnities for the present study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Area under curve from dosing time to last measurment (AUC (0-t)) for MD1003 | predose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264, 312 and 360 hours post-dose.
Area under curve from dosing tme to infinity (AUC(0-∞)) for MD1003 | predose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264, 312 and 360 hours post-dose.
Maximum plasma drug concentration (Cmax) for MD1003 | predose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264, 312 and 360 hours post-dose.
Measurement of concentration of MD1003 | predose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264, 312 and 360 hours post-dose.
Measurement of concentration of Bisnorbiotin | predose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264, 312 and 360 hours post-dose.
Measurement of concentration of Biotin sulfoxide | predose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264, 312 and 360 hours post-dose.

SECONDARY OUTCOMES:
Plasma pharmacokinetics: elimination half-life (t1/2) for MD1003 | predose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264, 312 and 360 hours post-dose.
Plasma pharmacokinetics: elimination half-life (t1/2) for Bisnorbiotin | predose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264, 312 and 360 hours post-dose.
  Blood samples will be collected
Plasma pharmacokinetics: elimination half-life (t1/2) for Biotin sulfoxide | predose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264, 312 and 360 hours post-dose.
  Blood samples will be collected
Plasma pharmacokinetics: time for maximum plasma concentration (tmax) for MD1003 | predose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264, 312 and 360 hours post-dose.
  Blood samples will be collected
Plasma pharmacokinetics: time for maximum plasma concentration (tmax) for Bisnorbiotin | predose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264, 312 and 360 hours post-dose.
  Blood samples will be collected
Plasma pharmacokinetics: time for maximum plasma concentration (tmax) for Biotin sulfoxide | predose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264, 312 and 360 hours post-dose.
  Blood samples will be collected
Plasma pharmacokinetics: elimination rate constant for MD1003 | predose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264, 312 and 360 hours post-dose.
  Blood samples will be collected
Plasma pharmacokinetics: elimination rate constant for Bisnorbiotin | predose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264, 312 and 360 hours post-dose.
  Blood samples will be collected
Plasma pharmacokinetics: elimination rate constant for Biotin sulfoxide | predose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264, 312 and 360 hours post-dose.
  Blood samples will be collected
Plasma pharmacokinetics:: Apparent volume of distribution for MD1003 | predose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264, 312 and 360 hours post-dose.
  Blood samples will be collected
Plasma pharmacokinetics:Aparrent clearance | predose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264, 312 and 360 hours post-dose.
  Blood samples will be collected
Plasma pharmacokinetics: Percentage of extrapolated AUC inf for MD1003 | predose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264, 312 and 360 hours post-dose.
  Blood samples will be collected
Plasma pharmacokinetics: Percentage of extrapolated AUC inf for Bisnorbiotin | predose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264, 312 and 360 hours post-dose.
  Blood samples will be collected
Plasma pharmacokinetics: Percentage of extrapolated AUC inf for Biotin sulfoxide | predose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264, 312 and 360 hours post-dose.
  Blood samples will be collected
Area under curve from dosing tme to infinity (AUC(0-∞)) for Bisnorbiotin | predose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264, 312 and 360 hours post-dose.
  Blood samples will be collected for the measurement of concentration for Bisnorbiotin
Area under curve from dosing tme to infinity (AUC(0-∞)) for Biotin sulfoxide | predose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264, 312 and 360 hours post-dose.
  Blood samples will be collected for the measurement of concentration for Biotin sulfoxide
Area under curve from dosing time to last measurement (AUC (0-t)) for Bisnorbiotin | predose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264, 312 and 360 hours post-dose.
  Blood samples will be collected for the measurement of concentration for Bisnorbiotin
Area under curve from dosing time to last measurement (AUC (0-t)) for Biotin sulfoxide | predose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264, 312 and 360 hours post-dose.
  Blood samples will be collected for the measurement of concentration for Biotin sulfoxide
Maximum plasma drug concentration (Cmax) for Bisnorbiotin | predose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264, 312 and 360 hours post-dose.
  Blood samples will be collected for the measurement for concentration for Bisnorbiotin
Maximum plasma drug concentration (Cmax) for Biotin sulfoxide | predose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264, 312 and 360 hours post-dose.
  Blood samples will be collected for the measurement of concentration for Biotin sulfoxide
Total amount excreted MD1003, Bisnorbiotin and Biotin sulfoxide urine over the time interval between t1 and t2 (Ae t1-t2) | predose to 168 hours post-dose
Total amount excreted MD1003, Bisnorbiotin and Biotin sulfoxide urine over the total time interval of urine collection (Ae0-t) | up to 168 hours post-dose
Renal calculated clairance | predose to 168 hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Yves Donazzolo, MD, Principal Investigator — Eurofins Optimed
Locations (5):
- Eurofins Optimed, Gières, France
- Hungary (4):
  - DRC Drug Research Center Ltd., Balatonfüred
  - Semmelweis University Faculty of Medicine, Budapest
  - University of Debrecen Medical and Health Center, Debrecen
  - Clinical Research Units Hungary Ltd., Miskolc